CLINICAL TRIAL: NCT01875185
Title: Hormones Inflammation and Thrombosis
Acronym: HIT2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funds for specimen management and data analysis
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00079522
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Acute Coronary Syndrome; Thrombosis
Keywords: acute coronary syndrome; clotting; hormones; women
MeSH Terms: conditions — Acute Coronary Syndrome; Thrombosis | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aspirin (Experimental): The patients are given aspirin 81 mg orally for 7 days.
  Interventions: Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Aspirin 81 mg — Aspirin 81 mg orally daily for 7 days
  Other Names: ASP

SUMMARY:
The investigators are attempting to determine if the response to aspirin in women is related to the level of estrogen and progesterone that a woman has.

DETAILED DESCRIPTION:
Thrombosis plays a significant role in both acute coronary syndromes (ACS) and early saphenous vein graft (SVG) failure. Women with coronary heart disease have higher levels of the inflammatory mediator thromboxane, which is produced by platelets, monocytes, macrophages and the endothelium. Data show that higher levels of urinary thromboxane (UTXB2) are associated with SVG failure 6 months after Coronary Artery Bypass Graft (CABG). Women in the study cohort had higher levels of UTXB2 and higher odds of graft failure when compared to men. The elevated urinary thromboxane seen in the women in our study cohort may represent a marker and/or an etiology of thrombosis.

Are the levels of UTXB2 higher in women due to hormonal differences? In a prior pilot study we investigated whether hormonal levels are associated with changes in urinary thromboxane. We looked at hormonal and urinary thromboxane levels in 48 postmenopausal and 52 premenopausal women. We found that postmenopausal women had higher levels of UTXB2 than did premenopausal women (2495 vs. 2299, p=.02) and that in premenopausal women a higher estrogen/progesterone ratio was associated with the highest levels of urinary thromboxane.

The goal of the current study is to measure the response to seven days of aspirin administration as it relates to urinary thromboxane levels in pre and post-menopausal women. With this study we will be able to examine the change in UTXB2 comparing the premenopausal to post menopausal women. We will also be able to see if the change in UTXB2 in response to aspirin is affected by hormone levels in the premenopausal women. Lastly this study will provide reference data for more far-reaching studies exploring how global changes in hormonal balance (as seen in pregnancy or menopause) or in the level of inflammation (as seen in aging or with Coronary Artery Disease (CAD) risk factors), affect UTXB2 and platelet hyperreactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 18-80
2. Signed informed consent.

Exclusion Criteria:

1. History of CAD, Cerebrovascular Accident (CVA) or Peripheral Artery Disease (PAD),
2. On chronic aspirin therapy,
3. On chronic NSAID therapy.
4. Chronic anticoagulation with coumadin,
5. Known thrombocytopenia (Platelet count < 100,000),
6. Pregnancy (self-report),
7. Currently on any type of contraceptive or hormone replacement therapy,
8. Hysterectomy and/or oophorectomy.
9. Recent GI bleeding
10. Bleeding diathesis
11. Chronic Systemic Infection

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhondalyn McLean, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Premenopausal; Postmenopausal: Aspirin 81 mg PO daily x 7 days
Period: Overall Study
Arm/Group | Premenopausal | Postmenopausal
Started | 52 | 48
Completed | 0 | 0
Not Completed | 52 | 48
Not completed — study was terminated | 52 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Premenopausal | Postmenopausal | Total
Number analyzed (Participants) | 52 | 48 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 0 | 52
  >=65 years | 0 | 48 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 48 | 100

OUTCOME MEASURES:

1. Primary Outcome: Level of Urinary Thromboxane (UTXB2) in pg/mg Creatinine
Description: Urinary thromboxane (pg/mg creatinine) will be measured in premenopausal and postmenopausal women at baseline and then after taking on aspirin for 7 days.
Time Frame: Baseline
Population: Data was only collected at baseline. The study was terminated prior to initiation of intervention (Aspirin) and therefore no follow-up data was collected to calculate the change from baseline.
Measure: Median (Inter-Quartile Range); unit: pg/mg
Groups:
- Premenopausal: premenopausal Women in the cohort
- Postmenopausal: Postmenopausal Women in the cohort
Arm/Group | Premenopausal | Postmenopausal
Number analyzed (Participants) | 52 | 48
pg/mg | 2495 [1775 to 3053] | 2299 [1724 to 2687]

2. Primary Outcome: The Change in the Level of UTXB2 in pg/mg Creatinine: Estrogen and Progesterone
Description: Measurement of urinary thromboxane (pg/mg creatinine) in relation to estrogen to progesterone level in premenopausal women on aspirin for 7 days.
Time Frame: baseline to 7 days
Population: Data was only collected at baseline. The study was terminated prior to obtaining study data.
Arm/Group | Premenopausal | Postmenopausal
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Level of UTXB2 in pg/mg Creatinine
Description: Comparing premenopausal women to postmenopausal women, the level of urinary thromboxane (pg/mg creatinine) in response to aspirin
Time Frame: baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/mg
Groups:
- Premenopausal: Premenopausal females in the cohort Aspirin 81 mg PO daily x 7 days
- Postmenopausal: Postmenopausal females in the cohort Aspirin 81 mg PO daily x 7 days
Arm/Group | Premenopausal | Postmenopausal
Number analyzed (Participants) | 52 | 48
pg/mg | 2299 [1724 to 2687] | 2824 [2198 to 3252]

4. Secondary Outcome: Relative Change of UTXB2 in pg/mg Creatinine in Response to Aspirin
Description: as for outcome 3
Time Frame: change from baseline to 7 days
Population: No data was collected for this outcome measure, as the study was terminated prematurely
Arm/Group | Premenopausal | Postmenopausal
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Premenopausal | Postmenopausal
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/48
Other Adverse Events (participants affected / at risk) | 0/52 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes